CLINICAL TRIAL: NCT00282048
Title: Phase 2 Study Of AG-013736 In Patients With Refractory Metastatic Renal Cell Cancer
Brief Title: Study Of AG-013736 In Patients With Refractory Metastatic Renal Cell Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A4061023
Record Dates: First submitted 2006-01-23; First posted 2006-01-25 (Estimated); Results first posted 2012-04-03 (Estimated); Last update posted 2012-07-31 (Estimated); Status verified 2012-07

CONDITIONS: Kidney Neoplasms; Carcinoma, Renal Cell
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — Axitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AG-013736 (axitinib) (Experimental): AG-013736 single agent in continuous dosing until disease progression or unacceptable toxicity
  Interventions: Drug: AG-013736 (axitinib)

INTERVENTIONS:
Drug: AG-013736 (axitinib) — AG-013736 5 mg twice daily [bid] continuous dosing in 28 day cycles.

SUMMARY:
To determine the activity and response rate of AG-013736 in patients with advanced and refractory renal cell cancer, (patients who also failed on sorafenib-based therapy).

ELIGIBILITY:
Inclusion Criteria:

* RCC with metastases and nephrectomy
* failure of prior sorafenib-based therapy
* at least 1 target lesion that has not been irradiated
* adequate bone marrow, hepatic and renal function, > or equal to 18 years of age.

Exclusion Criteria:

* Gastrointestinal abnormalities
* current use or inability to avoid chronic antacid therapy
* current use or anticipated inability to avoid potent CYP3A4 inhibitors or CYP1A2 inducers
* active seizure disorder or evidence of brain metastases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2006-03; Primary Completion 2009-02 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (5):
- United States (5):
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, The Bronx, New York
  - Pfizer Investigational Site, Cleveland, Ohio
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- Axitinib: Axitinib (AG-013736) tablet 5 milligram (mg) orally twice daily (BID) for 4 consecutive weeks (28 days cycle) with no interval between cycles.
Period: Overall Study
Arm/Group | Axitinib
Started | 62
Completed | 0
Not Completed | 62
Not completed — Lack of Efficacy | 30
Not completed — Adverse Event | 22
Not completed — Withdrawal by Subject | 1
Not completed — Other | 8
Not completed — Ongoing | 1

BASELINE CHARACTERISTICS:
Arm/Group | Axitinib
Number analyzed (Participants) | 62
Age Continuous [Mean (Standard Deviation); unit: Years] | 57.9 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 42

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Objective Response (OR)
Description: Percentage of participants with OR based assessment of confirmed complete response (CR) or confirmed partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST). Confirmed responses are those that persist on repeat imaging study at least 4 weeks after initial documentation of responses. CR are defined as the disappearance of all lesions (target and/or non target). PR are those with at least 30 percent (%) decrease in the sum of the longest dimensions of the target lesions taking as a reference the baseline sum of longest dimensions.
Time Frame: Baseline to disease progression or discontinuation from study due to any cause, assessed every 8 weeks up to 152 weeks
Population: Intent-to-treat (ITT) population included all enrolled participants who received at least 1 dose of the study medication, had a baseline assessment of disease and had the correct histological cancer type.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Axitinib
Number analyzed (Participants) | 62
Percentage of Participants | 22.6 [12.9 to 35.0]

2. Secondary Outcome: Progression-free Survival (PFS)
Description: Time in days from start of study treatment to first documentation of objective tumor progression or death due to any cause. PFS was calculated as first event date minus the date of first dose of study medication plus 1. Tumor progression was determined from oncologic assessment data (where data meet the criteria for progressive disease [PD]), or from adverse event (AE) data (where the outcome was "Death").
Time Frame: Baseline until the date of first documented progression or death due to any cause, assessed every 8 weeks up to 152 weeks
Population: ITT population included all enrolled participants who received at least 1 dose of the study medication, had a baseline assessment of disease and had the correct histological cancer type.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Axitinib
Number analyzed (Participants) | 62
Days | 225 [203 to 334]

3. Secondary Outcome: Duration of Response (DR)
Description: Time in days from the first documentation of objective tumor response to objective tumor progression or death due to any cancer. Duration of tumor response was calculated as the date of the first documentation of objective tumor progression or death due to cancer minus the date of the first CR or PR that was subsequently confirmed plus 1. DR was calculated for the subgroup of participants with a confirmed objective tumor response.
Time Frame: Baseline to disease progression or discontinuation from study due to any cause, assessed every 8 weeks up to 152 weeks
Population: Subgroup of participants from the ITT population, with a confirmed objective tumor response (CR or PR).
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Axitinib
Number analyzed (Participants) | 14
Days | 531 [225 to NA] — The upper limit was not estimable because large number of participants were censored.

4. Secondary Outcome: Overall Survival (OS)
Description: Time in days from the start of study treatment to date of death due to any cause. OS was calculated as the death date minus the date of first dose of study medication plus 1. Death was determined from AE data (where outcome was death) or from follow-up contact data (where the participant current status was death). For participants who were alive, overall survival was censored at the last contact.
Time Frame: Baseline to death due to any cause or at least 1 year after the first dose for the last participant
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Axitinib
Number analyzed (Participants) | 62
Days | 412.5 [256.0 to 570.0]

5. Secondary Outcome: Functional Assessment of Cancer Therapy (FACT)-Kidney Symptom Index for Disease Cancer Related Symptoms (FKSI-DRS) Score
Description: FKSI-DRS is a subset of FKSI which is a questionnaire for FACT -Kidney Symptom Index used to assess Quality of Life (QoL)/participant-reported outcomes for participants diagnosed with renal cell cancer. The FKSI contained 15 questions and the FKSI-DRS consisted of 9 questions each ranging from 0 (not at all) to 4 (very much) so that FKSI-DRS ranged between 0-36. Since the questions could be reversed coded, as appropriate, before calculating FKSI-DRS, 0 and 36 could be considered the worst and best health states based on the 9 questions comprising FKSI-DRS.
Time Frame: Baseline (Day 1 of Cycle 1), Day 1 of all subsequent cycles up to Cycle 38 and follow up (28 days after last dose)
Population: ITT population included all enrolled participants who received at least 1 dose of the study medication, had a baseline assessment of disease and had the correct histological cancer type. 'n' is the number of participants who completed at least one question.
Measure: Mean (95% Confidence Interval); unit: Units on a Scale
Arm/Group | Axitinib
Number analyzed (Participants) | 62
Units on a Scale
  Baseline (n=62) | 28.94 [27.69 to 30.19]
  Day 1 (Cycle 2) (n=52) | 27.12 [25.76 to 28.47]
  Day 1 (Cycle 3) (n=46) | 27.11 [25.79 to 28.43]
  Day 1 (Cycle 4) (n=41) | 27.68 [26.21 to 29.16]
  Day 1 (Cycle 5) (n=39) | 27.94 [26.55 to 29.34]
  Day 1 (Cycle 6) (n=33) | 27.31 [25.52 to 29.11]
  Day 1 (Cycle 7) (n=32) | 28.56 [26.79 to 30.33]
  Day 1 (Cycle 8) (n=30) | 28.55 [26.58 to 30.53]
  Day 1 (Cycle 9) (n=27) | 28.75 [27.05 to 30.44]
  Day 1 (Cycle 10) (n=19) | 29.37 [27.40 to 31.34]
  Day 1 (Cycle 11) (n=17) | 29.35 [27.13 to 31.57]
  Day 1 (Cycle 12) (n=17) | 29.24 [26.67 to 31.80]
  Day 1 (Cycle 13) (n=16) | 30.41 [28.27 to 32.56]
  Day 1 (Cycle 14) (n=15) | 31.02 [29.56 to 32.47]
  Day 1 (Cycle 15) (n=14) | 30.29 [28.48 to 32.09]
  Day 1 (Cycle 16) (n=14) | 30.79 [28.88 to 32.70]
  Day 1 (Cycle 17) (n=13) | 31.46 [29.10 to 33.82]
  Day 1 (Cycle 18) (n=12) | 31.08 [29.20 to 32.97]
  Day 1 (Cycle 19) (n=9) | 29.44 [26.72 to 32.17]
  Day 1 (Cycle 20) (n=10) | 29.80 [27.87 to 31.73]
  Day 1 (Cycle 21) (n=11) | 29.91 [26.71 to 33.11]
  Day 1 (Cycle 22) (n=10) | 30.80 [27.88 to 33.72]
  Day 1 (Cycle 23) (n=9) | 30.22 [25.74 to 34.70]
  Day 1 (Cycle 24) (n=8) | 31.75 [28.76 to 34.74]
  Day 1 (Cycle 25) (n=7) | 31.14 [27.58 to 34.70]
  Day 1 (Cycle 26) (n=7) | 31.29 [27.76 to 34.82]
  Day 1 (Cycle 27) (n=7) | 32.00 [28.08 to 35.92]
  Day 1 (Cycle 28) (n=5) | 34.00 [31.37 to 36.63]
  Day 1 (Cycle 29) (n=6) | 33.83 [31.49 to 36.17]
  Day 1 (Cycle 30) (n=6) | 34.00 [30.82 to 37.18]
  Day 1 (Cycle 31) (n=4) | 33.75 [28.49 to 39.01]
  Day 1 (Cycle 32) (n=1) | 34.00 [NA to NA] — 95% Confidence interval (CI) was not estimable because only 1 participant was evaluable.
  Day 1 (Cycle 33) (n=1) | 34.00 [NA to NA] — 95% CI was not estimable because only 1 participant was evaluable.
  Day 1 (Cycle 34) (n=0) | NA [NA to NA] — Mean was not estimable because no participant was evaluable.
  Day 1 (Cycle 35) (n=1) | 33.00 [NA to NA] — 95% CI was not estimable because only 1 participant was evaluable.
  Day 1 (Cycle 36) (n=1) | 33.00 [NA to NA] — 95% CI was not estimable because only 1 participant was evaluable.
  Day 1 (Cycle 37) (n=1) | 29.00 [NA to NA] — 95% CI was not estimable because only 1 participant was evaluable.
  Day 1 (Cycle 38) (n=1) | 30.00 [NA to NA] — 95% CI was not estimable because only 1 participant was evaluable.
  at Follow Up (n=9) | 25.11 [20.64 to 29.58]

6. Secondary Outcome: Population Pharmacokinetics of Axitinib (AG-013736)
Description: Data for this outcome measure are not reported here because the analysis population includes participants who were not enrolled in this study. ClinicalTrials.gov is designed for reporting results from only those participants who were enrolled in the study and described in the Participant Flow and Baseline Characteristics modules.
Time Frame: Day 1 (Pre-dose), Day 29, Day 57 and then every 8 weeks until disease progression or discontinuation from study or up to 152 weeks
Reporting Status: Not Posted
Measure: Mean (Standard Deviation); unit: nanogram/milliliter (ng/mL)

7. Other Pre Specified Outcome: Functional Assessment of Cancer Therapy (FACT)-Kidney Symptom Index (FKSI) Score
Description: FKSI is a questionnaire for FACT-Kidney Symptom Index used to assess QoL/participant-reported outcomes for participants diagnosed with renal cell cancer. The FKSI contained 15 questions each ranging from 0 (not at all) to 4 (very much) so that FKSI ranged between 0-60 where higher scores reflects better functioning and fewer symptoms.
Time Frame: Baseline (Day 1 of Cycle 1), Day 1 of all subsequent cycles up to Cycle 38 and follow up (28 days after last dose)
Population: as for outcome 5
Measure: Mean (95% Confidence Interval); unit: Units on a Scale
Arm/Group | Axitinib
Number analyzed (Participants) | 62
Units on a Scale
  Baseline (n=62) | 44.84 [42.65 to 47.03]
  Day 1 (Cycle 2) (n=52) | 41.40 [39.13 to 43.67]
  Day 1 (Cycle 3) (n=46) | 41.62 [39.28 to 43.97]
  Day 1 (Cycle 4) (n=41) | 42.26 [39.55 to 44.97]
  Day 1 (Cycle 5) (n=39) | 42.35 [39.85 to 44.84]
  Day 1 (Cycle 6) (n=33) | 41.65 [38.82 to 44.49]
  Day 1 (Cycle 7) (n=32) | 43.77 [41.09 to 46.45]
  Day 1 (Cycle 8) (n=30) | 44.00 [40.75 to 47.25]
  Day 1 (Cycle 9) (n=27) | 44.80 [41.84 to 47.76]
  Day 1 (Cycle 10) (n=19) | 45.39 [41.82 to 48.95]
  Day 1 (Cycle 11) (n=17) | 44.14 [40.23 to 48.06]
  Day 1 (Cycle 12) (n=17) | 44.73 [40.79 to 48.67]
  Day 1 (Cycle 13) (n=16) | 46.13 [42.19 to 50.06]
  Day 1 (Cycle 14) (n=15) | 47.04 [43.94 to 50.14]
  Day 1 (Cycle 15) (n=14) | 45.93 [42.67 to 49.20]
  Day 1 (Cycle 16) (n=14) | 46.16 [41.96 to 50.36]
  Day 1 (Cycle 17) (n=13) | 48.14 [44.18 to 52.10]
  Day 1 (Cycle 18) (n=12) | 47.08 [42.43 to 51.72]
  Day 1 (Cycle 19) (n=9) | 44.98 [39.24 to 50.71]
  Day 1 (Cycle 20) (n=10) | 45.81 [41.41 to 50.20]
  Day 1 (Cycle 21) (n=11) | 47.02 [40.99 to 53.05]
  Day 1 (Cycle 22) (n=10) | 47.50 [42.06 to 52.94]
  Day 1 (Cycle 23) (n=9) | 46.30 [38.77 to 53.83]
  Day 1 (Cycle 24) (n=8) | 48.64 [42.38 to 54.91]
  Day 1 (Cycle 25) (n=7) | 49.11 [44.46 to 53.77]
  Day 1 (Cycle 26) (n=7) | 50.26 [45.32 to 55.19]
  Day 1 (Cycle 27) (n=7) | 49.82 [43.61 to 56.02]
  Day 1 (Cycle 28) (n=5) | 53.20 [46.55 to 59.85]
  Day 1 (Cycle 29) (n=6) | 52.67 [45.84 to 59.49]
  Day 1 (Cycle 30) (n=6) | 53.17 [46.26 to 60.08]
  Day 1 (Cycle 31) (n=4) | 53.00 [40.74 to 65.26]
  Day 1 (Cycle 32) (n=1) | 53.00 [NA to NA] — 95% CI was not estimable because only 1 participant was evaluable.
  Day 1 (Cycle 33) (n=1) | 51.00 [NA to NA] — 95% CI was not estimable because only 1 participant was evaluable.
  Day 1 (Cycle 34) (n=0) | NA [NA to NA] — 95% CI was not estimable because no participant was evaluable.
  Day 1 (Cycle 35) (n=1) | 51.00 [NA to NA] — 95% CI was not estimable because only 1 participant was evaluable.
  Day 1 (Cycle 36) (n=1) | 51.00 [NA to NA] — 95% CI was not estimable because only 1 participant was evaluable.
  Day 1 (Cycle 37) (n=1) | 45.00 [NA to NA] — 95% CI was not estimable because only 1 participant was evaluable.
  Day 1 (Cycle 38) (n=1) | 48.00 [NA to NA] — 95% CI was not estimable because only 1 participant was evaluable.
  At Follow Up (n=9) | 38.98 [32.46 to 45.49]

8. Other Pre Specified Outcome: Correlation of Area Under the Concentration-time Curve at Steady State (AUCss) With Confirmed Partial Response (PR)
Description: AUCss: pharmacokinetic parameter derived from plasma concentration versus time data using non-compartmental or population based analysis methods, computed as each participant's average total daily dose (accounting for dose reductions and any recorded missed doses) divided by population estimated posthoc individual apparent clearance (CL/F), i.e., AUCss = Daily Dose/(CL/F), where F refers to the oral bioavailability, and CL refers to the systemic clearance. PR: responses with at least 30% decrease in sum of longest dimensions of target lesions using baseline (pre-treatment) sum of longest dimensions as reference. Logistic regression with general linear model was applied to data of PR using AUCss; PR was correlated with AUCss as fold increase in odds of PR with increase in AUCss. Fold increase was calculated as exponent of product of logistic regression slope coefficient and unit change of AUCss.
Time Frame: Day 1 (Pre-dose), Day 29 and then every 8 weeks until disease progression or discontinuation from study or up to 152 weeks
Population: Participants for whom both Pharmacokinetic (PK) and PR data were available were included in analysis.
Measure: Number; unit: Ratio
Arm/Group | Axitinib
Number analyzed (Participants) | 14
Ratio
  Fold change per 1 ng*hr/mL: Cycle1 | 1.0028
  Fold change per 100 ng*hr/mL: Cycle1 | 1.3300

9. Other Pre Specified Outcome: Relationship of Area Under the Concentration-time Curve at Steady State (AUCss) With Progression-free Survival (PFS)
Description: AUCss is a pharmacokinetic parameter derived from plasma concentration versus time data using non-compartmental or population based analysis methods. PFS is median time from first dose of study treatment to the first documentation of objective tumor progression or to death due to any cause, whichever occurs first. Relationship of PFS versus AUCss was determined as median PFS in participants with high AUCss [AUCss greater than or equal to (>=) median AUCss] or low AUCss [AUCss less than (<) median AUCss].
Time Frame: Day 1 (Pre-dose), Day 29, and then every 8 weeks until disease progression or discontinuation from study or up to 152 weeks
Population: Participants for whom both PK and PFS data were available were included in analysis. 'n' signifies number of participants evaluable for the corresponding category.
Measure: Median (Full Range); unit: weeks
Arm/Group | Axitinib
Number analyzed (Participants) | 57
weeks
  PFS at Low AUCss: Cycle1 (n=28) | 31 [24 to 80]
  PFS at High AUCss: Cycle1 (n=29) | 39 [31 to NA] — Upper limit of range was not estimable due to insuffecient number of progression events.

10. Other Pre Specified Outcome: Relationship of Area Under the Concentration-time Curve at Steady State (AUCss) With Overall Survival (OS)
Description: AUCss is a pharmacokinetic parameter derived from plasma concentration versus time data using non-compartmental or population based analysis methods. OS is time in weeks from the start of study treatment to date of death due to any cause. Relationship of OS versus AUCss was determined as median OS in participants with high AUCss [AUCss >= median AUCss] or low AUCss [AUCss < median AUCss].
Time Frame: as for outcome 8
Population: Participants for whom both PK and OS data were available were included in analysis. 'n' signifies number of participants evaluable for the corresponding category.
Measure: Median (Full Range); unit: weeks
Arm/Group | Axitinib
Number analyzed (Participants) | 57
weeks
  OS at Low AUCss: Cycle1 (n=28) | 43 [36 to 72]
  OS at High AUCss: Cycle1 (n=29) | 88 [73 to NA] — Upper limit of range was not estimable due to insuffecient number of progression events.

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Axitinib
Serious Adverse Events (participants affected / at risk) | 39/62
Other Adverse Events (participants affected / at risk) | 62/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Axitinib (N=62)
Atrial fibrillation (Cardiac disorders) | 1
Atrial tachycardia (Cardiac disorders) | 1
Bradycardia (Cardiac disorders) | 1
Bundle branch block left (Cardiac disorders) | 1
Cardiac disorder (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 2
Left ventricular dysfunction (Cardiac disorders) | 1
Myocardial ischaemia (Cardiac disorders) | 2
Tachycardia (Cardiac disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 5
Abdominal pain upper (Gastrointestinal disorders) | 1
Diverticulum (Gastrointestinal disorders) | 1
Gastrointestinal perforation (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Large intestine perforation (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 4
Chest pain (General disorders) | 1
Death (General disorders) | 1
Disease progression (General disorders) | 4
Fatigue (General disorders) | 2
Oedema peripheral (General disorders) | 1
Hepatorenal syndrome (Hepatobiliary disorders) | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1
Jaundice (Hepatobiliary disorders) | 1
Cholecystitis infective (Infections and infestations) | 1
Peritoneal infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Wound infection (Infections and infestations) | 1
Wound complication (Injury, poisoning and procedural complications) | 1
Blood alkaline phosphatase increased (Investigations) | 1
Blood creatinine increased (Investigations) | 1
Lipase increased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 6
Hypercalcaemia (Metabolism and nutrition disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2
Ataxia (Nervous system disorders) | 1
Cerebral haemorrhage (Nervous system disorders) | 2
Convulsion (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Lethargy (Nervous system disorders) | 2
Syncope (Nervous system disorders) | 2
Agitation (Psychiatric disorders) | 1
Confusional state (Psychiatric disorders) | 2
Mental status changes (Psychiatric disorders) | 1
Anuria (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Embolism arterial (Vascular disorders) | 1
Hypertension (Vascular disorders) | 3
Hypotension (Vascular disorders) | 5
Thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Axitinib (N=62)
Anaemia (Blood and lymphatic system disorders) | 3
Polycythaemia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 3
Left ventricular hypertrophy (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 2
Ventricular hypokinesia (Cardiac disorders) | 1
Hypoacusis (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Hypothyroidism (Endocrine disorders) | 11
Blindness (Eye disorders) | 1
Conjunctival haemorrhage (Eye disorders) | 1
Dry eye (Eye disorders) | 1
Eye pruritus (Eye disorders) | 1
Lacrimation increased (Eye disorders) | 1
Ocular hyperaemia (Eye disorders) | 1
Scleral haemorrhage (Eye disorders) | 1
Vitreous floaters (Eye disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 4
Abdominal pain (Gastrointestinal disorders) | 11
Abdominal pain lower (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 3
Anorectal discomfort (Gastrointestinal disorders) | 1
Cheilitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 16
Diarrhoea (Gastrointestinal disorders) | 38
Dry mouth (Gastrointestinal disorders) | 5
Dyspepsia (Gastrointestinal disorders) | 12
Dysphagia (Gastrointestinal disorders) | 2
Erosive oesophagitis (Gastrointestinal disorders) | 1
Eructation (Gastrointestinal disorders) | 4
Flatulence (Gastrointestinal disorders) | 5
Gastritis (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3
Gingivitis (Gastrointestinal disorders) | 1
Glossodynia (Gastrointestinal disorders) | 3
Haematochezia (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 2
Impaired gastric emptying (Gastrointestinal disorders) | 1
Large intestinal ulcer (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 27
Oral pain (Gastrointestinal disorders) | 7
Proctalgia (Gastrointestinal disorders) | 3
Rectal fissure (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 3
Stomatitis (Gastrointestinal disorders) | 11
Tongue ulceration (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 19
Asthenia (General disorders) | 1
Axillary pain (General disorders) | 1
Chest pain (General disorders) | 6
Chills (General disorders) | 7
Fatigue (General disorders) | 47
Hypothermia (General disorders) | 1
Impaired healing (General disorders) | 1
Influenza like illness (General disorders) | 1
Mucosal inflammation (General disorders) | 21
Non-cardiac chest pain (General disorders) | 1
Oedema peripheral (General disorders) | 11
Pain (General disorders) | 7
Pyrexia (General disorders) | 9
Suprapubic pain (General disorders) | 1
Temperature intolerance (General disorders) | 2
Bile duct obstruction (Hepatobiliary disorders) | 1
Hypersensitivity (Immune system disorders) | 3
Seasonal allergy (Immune system disorders) | 1
Abscess (Infections and infestations) | 1
Bacteraemia (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 2
Candidiasis (Infections and infestations) | 1
Ear infection (Infections and infestations) | 1
Folliculitis (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Localised infection (Infections and infestations) | 1
Oral candidiasis (Infections and infestations) | 1
Oral fungal infection (Infections and infestations) | 1
Oral infection (Infections and infestations) | 2
Pharyngitis (Infections and infestations) | 5
Pneumonia (Infections and infestations) | 4
Rhinitis (Infections and infestations) | 4
Septic shock (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 5
Tinea pedis (Infections and infestations) | 1
Tooth abscess (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 4
Urinary tract infection (Infections and infestations) | 8
Vaginal infection (Infections and infestations) | 1
Vulvovaginal mycotic infection (Infections and infestations) | 3
Wound infection (Infections and infestations) | 1
Contusion (Injury, poisoning and procedural complications) | 2
Gastrointestinal injury (Injury, poisoning and procedural complications) | 1
Procedural pain (Injury, poisoning and procedural complications) | 1
Splinter (Injury, poisoning and procedural complications) | 1
Activated partial thromboplastin time prolonged (Investigations) | 1
Alanine aminotransferase (Investigations) | 1
Alanine aminotransferase increased (Investigations) | 2
Aspartate aminotransferase (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 3
Blood alkaline phosphatase increased (Investigations) | 1
Blood amylase increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 1
Blood cholesterol increased (Investigations) | 1
Blood creatine increased (Investigations) | 2
Blood creatinine increased (Investigations) | 4
Blood lactate dehydrogenase increased (Investigations) | 1
Blood triglycerides increased (Investigations) | 1
Breath sounds abnormal (Investigations) | 1
International normalised ratio (Investigations) | 1
International normalised ratio increased (Investigations) | 2
Lipase increased (Investigations) | 1
Urobilinogen urine increased (Investigations) | 1
Weight decreased (Investigations) | 19
Decreased appetite (Metabolism and nutrition disorders) | 33
Dehydration (Metabolism and nutrition disorders) | 8
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hyperlipasaemia (Metabolism and nutrition disorders) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 16
Arthritis (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 8
Bone pain (Musculoskeletal and connective tissue disorders) | 6
Flank pain (Musculoskeletal and connective tissue disorders) | 2
Groin pain (Musculoskeletal and connective tissue disorders) | 2
Joint swelling (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 4
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 11
Neck pain (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 13
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1
Pubic pain (Musculoskeletal and connective tissue disorders) | 1
Ageusia (Nervous system disorders) | 1
Aphonia (Nervous system disorders) | 1
Balance disorder (Nervous system disorders) | 1
Brain mass (Nervous system disorders) | 1
Cognitive disorder (Nervous system disorders) | 1
Convulsion (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 11
Dysgeusia (Nervous system disorders) | 14
Extrapyramidal disorder (Nervous system disorders) | 1
Headache (Nervous system disorders) | 16
Hyperaesthesia (Nervous system disorders) | 2
Hypoaesthesia (Nervous system disorders) | 1
Neuropathy peripheral (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 6
Peripheral sensory neuropathy (Nervous system disorders) | 2
Peroneal nerve palsy (Nervous system disorders) | 2
Sciatica (Nervous system disorders) | 3
Tremor (Nervous system disorders) | 2
Anxiety (Psychiatric disorders) | 6
Confusional state (Psychiatric disorders) | 3
Depression (Psychiatric disorders) | 10
Disorientation (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 6
Bladder spasm (Renal and urinary disorders) | 1
Dysuria (Renal and urinary disorders) | 3
Glycosuria (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Micturition urgency (Renal and urinary disorders) | 2
Nocturia (Renal and urinary disorders) | 1
Pollakiuria (Renal and urinary disorders) | 3
Proteinuria (Renal and urinary disorders) | 8
Renal failure (Renal and urinary disorders) | 1
Urinary hesitation (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Breast oedema (Reproductive system and breast disorders) | 1
Erectile dysfunction (Reproductive system and breast disorders) | 1
Genital rash (Reproductive system and breast disorders) | 1
Scrotal disorder (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 17
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 23
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 21
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 10
Hiccups (Respiratory, thoracic and mediastinal disorders) | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 5
Dry skin (Skin and subcutaneous tissue disorders) | 9
Erythema (Skin and subcutaneous tissue disorders) | 4
Hair texture abnormal (Skin and subcutaneous tissue disorders) | 2
Hidradenitis (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 4
Nail discolouration (Skin and subcutaneous tissue disorders) | 1
Night sweats (Skin and subcutaneous tissue disorders) | 4
Pain of skin (Skin and subcutaneous tissue disorders) | 2
Palmar erythema (Skin and subcutaneous tissue disorders) | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 21
Petechiae (Skin and subcutaneous tissue disorders) | 1
Plantar erythema (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 4
Psoriasis (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Rosacea (Skin and subcutaneous tissue disorders) | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 2
Skin reaction (Skin and subcutaneous tissue disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 2
Swelling face (Skin and subcutaneous tissue disorders) | 1
Wound drainage (Surgical and medical procedures) | 1
Flushing (Vascular disorders) | 5
Haemorrhage (Vascular disorders) | 1
Hot flush (Vascular disorders) | 1
Hypertension (Vascular disorders) | 26
Hypotension (Vascular disorders) | 7
Thrombosis (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
Population pharmacokinetics was not presented, as the data was not available for the single study and data of other axitinib (AG-013736) Phase 2 studies would be pooled together in a separate report.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.